CLINICAL TRIAL: NCT01242423
Title: Accelerated Healing of Second Degree Burns and the Effect of Musculoskeletal Shockwave Therapy on the Recovery of Skin Graft Donor Sites
Brief Title: Healing of Burns and the Effect of Shockwave Therapy on the Recovery of Skin Grafts
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Unfallkrankenhaus Berlin (Other)
Responsible Party: Christian Ottoman, Unfallkrankenhaus Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA1/160/06
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Burn Wound and Skin Graft Healing
Keywords: musculoskeletal shockwave therapy
MeSH Terms: conditions — Burns | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- superficial 2nd degree burn (Experimental): Group A (n=50): Consent-capable male and female patients between ≥18 and ≤80 years of age who have sustained a superficial 2nd degree burn on ≥1% and ≤30% of the surface of the body.
  Interventions: Device: extracorporeal shockwave therapy
- deep 2nd degree burn (Experimental): Group B (n=50): Consent-capable male and female patients between ≥18 and ≤80 years of age who have sustained a deep 2nd degree burn on ≥1% and ≤30% of the surface of the body.
  Interventions: Device: extracorporeal shockwave therapy
- skin excision for the purpose of a skin graft (Experimental): Group C (n=50): Consent-capable male and female patients between ≥18 and ≤80 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of BBS.
  Interventions: Device: extracorporeal shockwave therapy

INTERVENTIONS:
Device: extracorporeal shockwave therapy — ESWT is administered as a one-off treatment on the wound surfaces within 24 hours of a 2nd degree burn trauma and immediately after an intraoperative skin graft excision procedure. A defocused sound head is orthogradely applied to the burn wound or the donor site. 100 impulses/cm² is administered at 20 seconds per cm². The defocused sound head is placed on the wound along with a sterile gel (Lavaseptgel®, Octenidingel®) and a sterile protection foil. The shockwaves deployed are not at an energy density that is painful. This single application of ESWT is followed by routine dressing using Mepitel® in combination with Polyhexanid/Octenidin®.
  Other Names: ESWT

SUMMARY:
The study is to review whether musculoskeletal shockwave therapy (ESWT) can speed up the healing of second-degree burns as well as skin-graft donor sites.

In both cases, the primary hypothesis is the shortened period leading up to the complete healing of the wound (reepithelization).

The secondary hypothesis in the course of the study assesses:

the rare manifestation of undesirable local events (e.g. reddening, swelling, hematoma).

DETAILED DESCRIPTION:
ESWT is administered as a one-off treatment on the wound surfaces within 24 hours of a 2nd degree burn trauma and immediately after an intraoperative skin graft excision procedure. A defocused sound head is orthogradely applied to the burn wound or the donor site. 100 impulses/cm² is administered at 20 seconds per cm². The defocused sound head is placed on the wound along with a sterile gel (Lavaseptgel®, Octenidingel®) and a sterile protection foil. The shockwaves deployed are not at an energy density that is painful. This single application of ESWT is followed by routine dressing using Mepitel® in combination with Polyhexanid/Octenidin®.

ELIGIBILITY:
Inclusion Criteria:

Group A (n=50): Consent-capable male and female patients between ≥18 and ≤80 years of age who have sustained a superficial 2nd degree burn on ≥1% and ≤30% of the surface of the body.

Group B (n=50): Consent-capable male and female patients between ≥18 and ≤80 years of age who have sustained a deep 2nd degree burn on ≥1% and ≤30% of the surface of the body.

Group C (n=50): Consent-capable male and female patients between ≥18 and ≤80 years of age who require a skin excision for the purpose of a skin graft. The minimal size of the skin-graft donor site must not be less than 1% of BBS.

Exclusion Criteria:

General exclusion criteria

1. pregnancy
2. below 18 or above 80 years of age
3. burns requiring artificial respiration, since consent for the study participation is unobtainable
4. extent of burns ≤1% to ≥30% of the body surface

Anamnestic exclusion criteria

1. diabetes mellitus requiring insulin
2. dialysis-dependent
3. ongoing chemotherapy treatment
4. drug abuse
5. systemic skin diseases
6. systemic and local cortisone therapy

Local exclusion criteria

Excluded from the study are those with burns in the regions:

1. head, face, neck
2. proximal ventral and dorsal thorax

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The period leading up to the complete healing of the wound (reepithelization).

SECONDARY OUTCOMES:
Manifestation of undesirable local events (e.g. reddening, swelling, hematoma).

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hartmann, MD, Principal Investigator — Unfallkrankenhaus Berlin
Locations (1):
- Unfallkrankenhaus Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Ottomann C, Stojadinovic A, Lavin PT, Gannon FH, Heggeness MH, Thiele R, Schaden W, Hartmann B. Prospective randomized phase II Trial of accelerated reepithelialization of superficial second-degree burn wounds using extracorporeal shock wave therapy. Ann Surg. 2012 Jan;255(1):23-9. doi: 10.1097/SLA.0b013e318227b3c0. PMID 21775883